CLINICAL TRIAL: NCT02545153
Title: Randomised Controlled Trial of Fibrin Sealant to Prevent Bile Leakage After Cholangiotomy
Brief Title: Fibrin Sealant for Cholangiotomy Closure Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lasarettet i Enköping (Other)
Responsible Party: Principal Investigator, BAHMAN DARKAHI, MD, Lasarettet i Enköping
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: glue 55 galla
Record Dates: First submitted 2012-10-10; First posted 2015-09-09 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Common Bile Duct Gall Stones; Infection; Bile Leak
MeSH Terms: conditions — Gallstones; Infections | interventions — Fibrin Tissue Adhesive; Aprotinin; Fibrinogen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fibrin sealant (Active Comparator): Tisseel, Baxter (Aprotinin and Fibrinogen)
  Interventions: Drug: Tisseel, Baxter (Aprotinin and Fibrinogen)
- Control (Placebo Comparator): Suturing the incision without fibrin glue
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Tisseel, Baxter (Aprotinin and Fibrinogen) — After introducton of t tube and closure of the incision with running sutures, fibrin sealant is applied on the incision.
  Other Names: Closing the incision with fibrin sealant
  Arms: Fibrin sealant
Drug: Control — No fibrin sealant applied
  Other Names: Closing the incision without fibrin sealant
  Arms: Control

SUMMARY:
Bile leak reduction from the common bile duct, as a result of glue appliance after cholangiotomy.

DETAILED DESCRIPTION:
Laparoscopic common bile duct exploration is a way of dealing with common bile duct stones that has gained increasing acceptance. Following a cholangiotomy there is, however, the risk of bile leakage from the incision.

A way of avoiding leakage following cholangiotomy may be to apply fibrin sealant on the cholangiotomy.

The present study is based on patients undergoing laparoscopic cholecystectomy at the department of surgery, Enköping hospital, Sweden. The patients are informed about the study prior to the procedure. Cholangiography is performed routinely. In case common bile duct stones are encountered on the cholangiography, an incision is made in the common bile duct and the stones are extracted. After the stone extraction, a t tube is introduced into the cholangiotomy and the incision is closed with running Vicryl sutures.

When the cholangiotomy has been closed, the randomisation is performed with a sealed envelope system. If the patient is randomised to fibrin sealant, this is applied on the cholangiotomy. A passive drain is introduced before the abdomen is closed.

Postoperatively, the amount of bile in the passive drain is measured by an observer randomised to the allocation.

If the amount of bile in the drain does not exceed 100 ml three days postoperatively, a secondary cholangiography is performed through the t tube. If the contrast passes to the duodenum and no contrast leakage is seen, the t tube is withdrawn.

All postoperative complications are registered according to the Clavien-Dindo system.

ELIGIBILITY:
Inclusion Criteria:

* Gallbladder disease

Exclusion Criteria:

* Cancer/Tumor

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative biliary leakage | From the the day of surgery until discharge and/or removal of abdominal drain, up to two weeks
  The amount of bile in the drain is measured daily until it is withdrawn

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Sandblom, Assoc Prof, Principal Investigator — Karolinska Institutet
Locations (1):
- Lasarettet i Enkoping, Enköping, Uppsala County, Sweden

REFERENCES:
- [Derived] Darkahi B, Norden T, Sandblom G. Fibrin Sealant for Prevention of Bile Leakage After Laparoscopic Common Bile Duct Incision: Outcome of a Randomized Controlled Trial. J Laparoendosc Adv Surg Tech A. 2022 Feb;32(2):171-175. doi: 10.1089/lap.2020.0404. Epub 2021 Jun 14. PMID 34129409